CLINICAL TRIAL: NCT07211932
Title: Efficacy of Tofacitinib in Patients With Juvenile Idiopathic Arthritis: A Study Based on Real-world Clinical Practice Data.
Brief Title: Tofacitinib in Juvenile Idiopathic Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-78
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
Keywords: Arthritis, Juvenile; tofacitinib [Supplementary Concept]; Janus Kinase Inhibitors
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tofacitinib: Patients affected by JIA and treated with tofacitinib
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Patients received tofacitinib for the treatment of juvenile idiopathic arthritis (JIA).

SUMMARY:
This study aims to evaluate, using real-world clinical practice data, the efficacy of tofacitinib in improving the clinical control of juvenile idiopathic arthritis (JIA) after 12 months of treatment.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of juvenile idiopathic arthritis (JIA) documented in the medical record by the treating rheumatologist.

Documentation in the medical record of the medical indication for tofacitinib treatment, with a diagnostic justification related to JIA.

Age under 18 years at the time of the treatment indication with tofacitinib.

Exclusion criteria:

Participants diagnosed with any of the following conditions:

Reactive arthritis

Arthritis associated with inflammatory bowel disease

Arthritis associated with another autoimmune disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with JIA
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
JADAS-10 | Baseline and 12 months
  Change in the Juvenile Arthritis Disease Activity Score (JADAS-10) score at 12 months of treatment with tofacitinib. Range score: 0 to 10, the less score the better

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Sant Joan de Déu Barcelona, Barcelona, Barcelona
  - Corporació Sanitària Parc Taulí de Sabadell, Sabadell, Barcelona
  - Hospital de Vilafranca, Vilafranca del Penedès, Barceona

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.